CLINICAL TRIAL: NCT07327203
Title: Video-based Guided Self Help Dialectical Behavior Therapy for Binge Eating Disorder
Acronym: VIDEO-DBT-GSH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Táki Athanássios Cordás, Coordinator, Eating Disorders Program, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 88641125.1.0000.006
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Binge Eating Disorder
Keywords: BED; DBT; Dialectical Behavior Therapy; Guided Self-Help; Video-based intervention; DBT-BED; DBTgsh
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Beds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-based DBTgsh for BED (Experimental): Participants assigned to the experimental group will receive a 13-week guided self-help intervention based on Dialectical Behavior Therapy for Binge Eating Disorder (DBT-BED), delivered through weekly video lessons. The content is structured into three progressive modules covering core DBT skills: (1) mindfulness, (2) emotion regulation, and (3) distress tolerance. The video lessons will be adapted from the Portuguese version of The DBT Solution for Emotional Eating (Safer, Adler & Masson, 2020).
  In addition to the video content, participants will have access to six brief online sessions with a psychologist (30 minutes each), conducted via videoconference. These sessions will be distributed as follows: two in the first two weeks, three biweekly, and one at the end of the treatment.
  Interventions: Behavioral: Experimental: Video-based DBTgsh for BED
- Traditional DBTgsh for BED (text-based model) (Active Comparator): Participants in the control group will receive the traditional guided self-help version of DBT-BED, using the guided self-help manual of The DBT Solution for Emotional Eating in the Portuguese version (Safer, Adler & Masson, 2020). Participants will be instructed to read one chapter per week over the 13-week treatment period. The content covers the same three core DBT modules: mindfulness skills, emotion regulation, and distress tolerance. As in the experimental group, participants will also participate in six online sessions with a psychologist (30 minutes each), following the same time schedule. These sessions will have the same objectives as those in the experimental group.
  Interventions: Behavioral: Traditional DBTgsh for BED (text-based model)

INTERVENTIONS:
Behavioral: Experimental: Video-based DBTgsh for BED — This is a guided self-help behavioral intervention based on Dialectical Behavior Therapy for Binge Eating Disorder (DBT-BED), delivered through weekly pre-recorded video lessons over 13 weeks. The intervention covers three core DBT skill modules-mindfulness, emotion regulation, and distress tolerance-and is supported by six brief 30-minute individual online guidance sessions with a psychologist to enhance adherence, clarify content, and support skill application.
  Arms: Video-based DBTgsh for BED
Behavioral: Traditional DBTgsh for BED (text-based model) — This is a guided self-help behavioral intervention based on Dialectical Behavior Therapy for Binge Eating Disorder (DBT-BED), delivered through weekly chapter readings from a structured manual over 13 weeks. The intervention covers the same three core DBT skill modules-mindfulness, emotion regulation, and distress tolerance-and is supported by six brief 30-minute individual online guidance sessions with a psychologist to enhance adherence, clarify content, and support skill application.
  Arms: Traditional DBTgsh for BED (text-based model)

SUMMARY:
Dialectical Behavior Therapy (DBT) is an effective treatment for eating disorders, showing promising remission rates for Binge Eating Disorder (BED) in both standard and guided self-help formats. Traditional guided self-help models typically combine weekly chapter readings with a limited number of brief therapist meetings. However, the requirement of weekly book readings can be particularly challenging for individuals with BED, who often exhibit impulsive personality traits, psychiatric comorbidities, and weight-related health problems.

This study was developed to test a version of guided self-help DBT-BED delivered through video lessons instead of text. This randomized clinical trial will be conducted at the Eating Disorders Program of the Institute of Psychiatry, Hospital das Clínicas, Faculty of Medicine, University of São Paulo (AMBULIM IPq HC FMUSP), Brazil. Eighty adults with BED will be randomized to either an experimental group (weekly video lessons) or a control group (weekly text-based readings).

Both groups will undergo a 13-week intervention, including six brief 30-minute online guidance sessions with a psychologist. The primary outcome will be full remission from binge eating episodes at the end of treatment and at the 3-month follow-up. Secondary outcomes will include changes in eating disorder psychopathology, emotion regulation, quality of life, self-esteem, and dropout rates. Statistical analyses will follow the intention-to-treat principle.

DETAILED DESCRIPTION:
The aim of this randomized controlled trial is to compare the efficacy of a video-based adaptation of guided self-help Dialectical Behavior Therapy for adults with Binge Eating Disorder (BED) with the traditional text-based guided self-help format. The study focuses on clinical remission of binge eating episodes, treatment adherence, and maintenance of therapeutic effects over time.

Eighty adults diagnosed with BED will be recruited through the Eating Disorders Program of the Institute of Psychiatry at the Hospital das Clínicas, Faculty of Medicine, University of São Paulo (AMBULIM IPq HC FMUSP), Brazil. Participants will be randomly assigned to one of two intervention groups. The experimental group will receive the content of the guided self-help DBT-BED manual delivered through weekly video lessons based on the book chapters. The control group will receive the same content in a traditional text-based guided self-help format, following the same weekly structure.

Both groups will participate in six brief individual online guidance sessions with a psychologist, each lasting approximately 30 minutes. These sessions are intended to support treatment engagement, clarify intervention content, address treatment-interfering behaviors, promote generalization of DBT skills, and enhance motivation throughout the intervention.

Assessments will be conducted at baseline, at the end of the intervention period, and at a 3-month follow-up. The primary outcome of the study will be complete remission of binge eating episodes at post-treatment and follow-up. Secondary outcomes will include changes in eating disorder psychopathology, emotional regulation, quality of life, self-esteem, and treatment dropout rates.

The study is scheduled to begin in February 2026, with anticipated completion in December 2026.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with binge eating disorder according to the DSM-5-TR.
* Access to a device with a camera, microphone, and internet connection.
* Minimum ability to read and write in Portuguese.
* Availability of 1 hour per week to read or watch treatment-related content.
* Participants with psychiatric comorbidities must be on a stable medication regimen for at least two months prior to enrollment in the study.

Exclusion Criteria:

* Individuals with anorexia nervosa or bulimia nervosa.
* Individuals with unstable psychiatric comorbidities (exclusion will apply to individuals who have experienced an acute psychiatric exacerbation requiring additional treatment or medical hospitalization.).
* Lack of time to read weekly chapters or watch the video lessons.
* Inability to access devices with a camera, microphone, and internet.
* Inability to attend six brief 30-minute videoconference sessions over the 13-week study period.
* Individuals at imminent risk to life (suicidal or self-harming behavior in the previous three months).
* Lack of minimum reading and writing skills.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-10-23 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q) | Pre-treatment (baseline), post-treatment at 13 weeks, and 3-month follow-up.
  Eating Disorder Examination Questionnaire (EDE-Q) is a self-report measure assessing the severity of eating disorder psychopathology, including binge eating-related symptoms. The global score is calculated as the mean of four subscales. Scores range from 0 to 6, with higher scores indicating greater eating disorder psychopathology.

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | Pre-treatment (baseline), post-treatment at 13 weeks, and 3-month follow-up.
  Difficulties in Emotion Regulation Scale (DERS) is a self-report measure assessing difficulties across multiple aspects of emotional regulation, including emotional awareness, acceptance of emotional responses, impulse control, and access to effective emotion regulation strategies. The total score is calculated as the sum of 36 items. Scores range from 36 to 180, with higher scores indicating greater difficulties in emotion regulation.
Short Form Health Survey (SF-36) | Pre-treatment (baseline), post-treatment at 13 weeks, and 3-month follow-up.
  Short Form Health Survey (SF-36) is a generic self-report questionnaire assessing health-related quality of life across multiple domains, including physical functioning, role limitations due to physical or emotional problems, bodily pain, vitality, social functioning, emotional well-being, and general health perception. Scores range from 0 to 100, with higher scores indicating better perceived health status and fewer functional limitations.
Rosenberg Self-Esteem Scale (RSES) | Pre-treatment (baseline), post-treatment at 13 weeks, and 3-month follow-up.
  Rosenberg Self-Esteem Scale (RSES) is a self-report instrument designed to assess global self-esteem, reflecting overall feelings of self-worth and self-acceptance. The scale consists of 10 items rated on a Likert-type format, with the total score calculated as the sum of all items. Scores range from 0 to 30, with higher scores indicating higher levels of self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Táki Cordas, Medical Coordinator, Study Director — Eating Disorders Program of the Psychiatry Institute, Hospital das Clínicas, Medical School, University of São Paulo (AMBULIM IPq HC FMUSP), Brazil.
Locations (1):
- AMBULIM IPq HC FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
At the time of registration, a decision regarding the sharing of individual participant data (IPD) has not yet been made. The research team will evaluate the feasibility of IPD sharing after study completion, considering ethical approvals, participant consent, data protection regulations, and institutional policies. Any future data sharing will be limited to de-identified data and will follow applicable legal and ethical requirements.

REFERENCES:
- [Background] Ben-Porath, D., Duthu, F., Luo, T., Gonidakis, F., Compte, E. J., & Wisniewski, L. (2020). Dialectical behavioral therapy: an update and review of the existing treatment models adapted for adults with eating disorders. Dialectical Behavior Therapy for Eating Disorders, 5-25. DOI: 10.1080/10640266.2020.1723371. Carter, J. C., Kenny, T. E., Singleton, C., Van Wijk, M., & Heath, O. (2020). Dialectical behavior therapy self-help for binge-eating disorder: A randomized controlled study. International Journal of Eating Disorders, 53(3), 451-460.Masson, P. C., von Ranson, K. M., Wallace, L. M., & Safer, D. L. (2013). A randomized wait-list controlled pilot study of dialectical behaviour therapy guided self-help for binge eating disorder. Behaviour research and therapy, 51(11), 723-728.Safer, D. L., Adler, S., & Masson, P. C. (2018). The DBT solution for emotional eating: A proven program to break the cycle of bingeing and out-of-control eating. Guilford Publications.